CLINICAL TRIAL: NCT06914596
Title: Randomized Controlled Clinical Trial To Assess The Safety and Effectiveness of A Periodontal Hydrogel Dressing (Emanate Perio PODS) On Wound Healing Post-Scaling and Root Planing
Brief Title: A Clinical Trial Comparing Overnight and 2x/Day for 30-minutes Use of the Emanate Perio PODS Post-SRP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGuire Institute (Industry)
Collaborators: Emanate Biomedical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EB2025-01
Record Dates: First submitted 2024-12-30; First posted 2025-04-06 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-03

CONDITIONS: Periodontitis (Stage 3)
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Randomized, examiner-blind, controlled, three-armed, parallel group, multi-site clinical trial comparing overnight and 2x/day for 30-minutes use of the Emanate Perio PODS post-SRP
Masking Description: At each study site, study roles will be designated such that the blinded examiner procedures will be separate from the clinicians conducting the other evaluations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Group A - Overnight PODS (Experimental): Overnight use of Emanate Perio PODS for 14 days post-SRP
  Interventions: Device: Emanate Perio PODS
- Group B - 2x/day PODS (Experimental): Emanate Perio PODS used 2x/day for 30 minutes for 14 days post-SRP
  Interventions: Device: Emanate Perio PODS
- Group C - Control (No Intervention): No treatment post-SRP (Control Group)

INTERVENTIONS:
Device: Emanate Perio PODS — Emanate Perio PODS used overnight for 14 days post-SRP
  Arms: Group A - Overnight PODS
Device: Emanate Perio PODS — Emanate Perio PODS used 2x/day for 30 minutes use
  Arms: Group B - 2x/day PODS

SUMMARY:
The goal of this clinical trial is to compare safety and to see if individuals with generalized stage III periodontitis that are given a periodontal hydrogel dressing on a wound healing after plaque and tartar have been removed from teeth have greater healing than individuals who are given no treatment after.

DETAILED DESCRIPTION:
Periodontitis can be considered a chronic wound, in which the barrier has been compromised allowing pathogenic bacteria to infiltrate the subgingival space.

In this study, the Emanate Perio PODS dressing is applied for 30 minutes and overnight immediately after toothbrushing and interdental cleaning to physically protect the healing periodontal pocket from pathogenic bacteria while the epithelium reestablishes itself; which usually takes between 15-30 minutes. By week four post SRP, the epithelium matures enough to withstand the mechanical forces and therefore the treatment can stop. It is hypothesized that during the initial phases of healing, i.e., day 1 to day 30, and in the absence of mechanical forces, the epithelium can protect the subgingival pocket, and Emanate Perio PODS dressing is only applied after toothbrushing and interdental cleaning when tissue is exposed to disruptive mechanical forces. The limited use of the device minimizes the burden of use on patients and aligns with recommended twice daily toothbrushing which can improve treatment adherence and compliance.

ELIGIBILITY:
Inclusion Criteria

1. Subjects will have read, understood, and signed an institutional review board (IRB) approved Informed Consent Form (ICF).
2. Subjects 22 to 75 years of age.
3. Generalized Stage III periodontitis with at least 8 teeth having interproximal clinical attachment level of ≥3 mm and a probing pocket depth of ≥5 mm and ≤7mm, distributed between the mandible and the maxilla, with at least 2 qualifying interproximal sites in each arch. Localized and not more than 6 sites with a PD of 8 mm is acceptable as long as the tooth with 8 mm pocket depth is not clinically diagnosed as hopeless tooth with suppuration or mobility Grade 3 or greater.5-7
4. Subjects have a minimum of 24 natural teeth with a minimum of 2 natural teeth per quadrant excluding third molars.
5. All supragingival accretions can be removed from below the height of contour of the tooth crown to allow for a comprehensive periodontal evaluation and accurate intraoral digital scan of both arches at screening.
6. Subjects agree to refrain from use of oral rinses or dentifrice with known antibacterial properties (e.g., Peridex®, Listerine®, Colgate Total®, Crest Pro-Health®, etc.).
7. Subjects agree to refrain from use of electric flossers or irrigation devices for the duration of the study.
8. Subjects can provide self-care (oral hygiene) without disabilities requiring assistance with daily oral hygiene measures.
9. Subjects are able and willing to follow study procedures and instructions

Exclusion Criteria:

1. Periodontal surgery, implant placement or SRP within 12 months prior to screening or a cleaning/prophylaxis six months prior to screening.
2. Presence of fixed or removable (e.g. Invisalign) orthodontic appliances.
3. Subject with an underlying medical condition which requires antibiotic prophylaxis prior to dental treatment.
4. Subjects with vesiculobullous processes or other similar chronic oral lesions / conditions resulting in gingival irritation, discomfort/pain, or erosions.
5. Subjects with soft or hard tissue tumor(s) of oral cavity.
6. Use of any smoked substances such as tobacco / cannabis including cigarettes, vape, cigars, or use of smokeless tobacco 30 days prior to screening and throughout the study.
7. Uncontrolled medical conditions (e.g., diabetes mellitus, hypertension, cancer).
8. Subjects who are lactating or pregnant or planning to become pregnant through their projected study duration.
9. Subjects taking medications known to affect gingival conditions. (e.g., hyperplasia).
10. Regular, prolonged use of oral antimicrobial rinses 30 days prior to screening or continued anticipated use through their projected study duration.
11. Use of systemic antibiotics 30 days prior to screening or anticipated during the trial period.
12. Subjects taking corticosteroids on a regular basis one week prior to baseline examination and throughout the duration of the study, including oral inhalers.
13. Subjects taking non-steroidal anti-inflammatory (NSAIDS) or other pain medication on a daily basis for more than 3 consecutive days beginning one week prior to the baseline examination and throughout the duration of the study. Subjects are allowed to take 81 mg/day aspirin and may use oral pain medication if needed in the first 48-hours post-SRP period.
14. Subjects taking anticoagulant medications such as warfarin or Plavix or Eliquis.
15. Subjects participating in other clinical studies involving therapeutic intervention (either medical or dental) within 30 days of Screening.
16. Subjects that are known to be hypersensitive to chlorhexidine gluconate, glycerin, polyvinyl alcohol or ethylene vinyl acetate.
17. Subjects, who in the opinion of the investigator, for any reason other than those listed above, will not be able to complete the study per protocol.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness on periodontal wound healing compared to control as evidenced by the presence/absence of gingival bleeding | 60 Days post non-surgical therapy
  Change in Bleeding on Marginal Probing (BOMP) over time at 60 Days post non-surgical therapy

SECONDARY OUTCOMES:
Effectiveness on periodontal wound healing compared to control | 60 Days post non-surgical therapy
  As evidenced by change in Modified Gingival Index (MGI)
Effectiveness on periodontal wound healing compared to control | 60 Days post non-surgical therapy
  As evidenced by change change in Pocket Depth (PD) over time in sites with baseline pockets >/=4mm

OTHER OUTCOMES:
Effectiveness on periodontal wound healing compared to the historical treatment effect of non-surgical therapy | 60 Days post non-surgical therapy
  Change in Pocket Depth (PD) over time in sites with baseline pockets >/=4mm at 60 days post non-surgical therapy
Feasibility of usage of the Emanate Perio PODS overnight group and the twice a day group | Day 14
  Feasibility will be characterized by compliance at Day 14 post non-surgical therapy
Feasibility of usage of the Emanate Perio PODS overnight group and the twice a day group | Pre-treatment, Day 14, Day 30
  Feasibility will be characterized by Dropout rate pre-treatment and at day 14 and Day 30
Feasibility of usage of the Emanate Perio PODS overnight group and the twice a day group | Pre-treatment, Day 14
  Feasibility will be characterized by mouthpiece fit and comfort as measured using the VAS at Day 0 and at Day 14 post non-surgical therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jarret Fass, Study Director — Emanate Biomedical
Locations (6):
- United States (6):
  - Shoreline Periodontics and Dental Implants, New London, Connecticut
  - Metro West Orthodontics & Periodontics, La Vista, Nebraska
  - Perio Health Professionals, Houston, Texas
  - Gulf Coast Periodontics, Victoria, Texas
  - Glazier Implants + Periodontics, Richmond, Virginia
  - Richardson, Overstreet, & White Ltd., Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No